CLINICAL TRIAL: NCT03532139
Title: Pilot Study of Rosuvastatin and Enoxaparin Thromboprophylaxis Following Ovarian Cancer Surgery (O-STAT Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Rushad Patell, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-067; 1R34HL135226-01 (NIH)
Record Dates: First submitted 2018-04-27; First posted 2018-05-22 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Enoxaparin; Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to Arm Enoxaparin and Arm Enoxaparin + Rosuvastatin, and those requesting no randomization willl be directly assigned to Arm Standard-of-care Thromboprophylaxis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Enoxaparin (Experimental): -Enoxaparin is administered subcutaneous daily
  Interventions: Drug: Enoxaparin
- Enoxaparin + Rosuvastatin (Experimental): * Enoxaparin is administered subcutaneous daily.
  * Rosuvastatin is administered daily orally starting on day 15
  Interventions: Drug: Enoxaparin; Drug: Enoxaparin + Rosuvastatin
- Thromboprophylaxis (Experimental): -Thromboprophylaxis is administered per clinician discretion
  Interventions: Other: Thromboprophylaxis

INTERVENTIONS:
Drug: Enoxaparin — Enoxaparin is used for prevention of blood clots following abdominal or orthopedic surgery and in medical patients with restricted mobility during acute illness
  Arms: Enoxaparin; Enoxaparin + Rosuvastatin
Drug: Enoxaparin + Rosuvastatin — Rosuvastatin is an anti-cholesterol medication that is FDA (the U.S. Food and Drug Administration) approved to lower cholesterol and reduce the risk of arterial blood clots. There is evidence that rosuvastatin can lower the risk of venous blood clots in healthy individuals
  Enoxaparin is used for prevention of blood clots following abdominal or orthopedic surgery and in medical patients with restricted mobility during acute illness
  Arms: Enoxaparin + Rosuvastatin
Other: Thromboprophylaxis — standard of care therapy
  Arms: Thromboprophylaxis

SUMMARY:
This research study is studying a combination of two drug interventions called rosuvastatin and enoxaparin as a possible preventative measure against developing venous blood clots (such deep vein thrombosis or pulmonary embolism). .

The drugs involved in this study are:

* Rosuvastatin, also known as Crestor
* Enoxaparin

DETAILED DESCRIPTION:
This is a randomized pilot trial to estimate the effect of rosuvastatin on levels of tissue factor bearing microparticles (TFMP) in patients undergoing surgery for presumed ovarian cancer (including primary peritoneal and fallopian tube carcinoma). Women will either be randomized to enoxaparin subcutaneously once daily (Arm A) or enoxaparin in combination with rosuvastatin (Arm B). Arm C will receive thromboprophylaxis according to standard of care and not be randomized. Levels of circulating TFMP will be assessed in all patients on Day 1 and following surgery (days 15, 30 and day 60). A bilateral lower extremity ultrasound will be performed on days 30 and 60 for all participants to estimate the rate of VTE in the 3 arms.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of ovarian, fallopian or primary peritoneal cancer (excluding borderline histologies). Preliminary pathology results based on frozen section findings are acceptable.
* The interval between pelvic or abdominal surgery and first dose of study treatment must be no more than 10 days.
* Age ≥ 18 years.
* ECOG performance status ≤2 (see Appendix A)
* Life expectancy of greater than 6 months
* Participants must have normal organ and marrow function as defined below:

  * Platelets ≥ 100,000/mcL
  * Total Bilirubin <1.5 mg/dL (or direct bilirubin <1.0 mg/dL)
  * AST(SGOT) ≤ 1.5 × institutional upper limit of normal
  * ALT(SGPT) ≤ 1.5 × institutional upper limit of normal
  * Creatinine < 1.5 mg/dL OR
  * Estimated creatinine clearance ≥60 mL/min/1.73 m2
* The effects of rosuvastatin on the developing human fetus are unknown. For this reason and because statins used in this trial are thought to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who are receiving any other investigational agents.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and increased risk of intracranial hemorrhage
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to enoxaparin or atorvastatin
* Active bleeding or high risk of bleeding (e.g. known acute gastrointestinal ulcer)
* History of heparin-induced thrombocytopenia.
* Any history of significant hemorrhage (requiring hospitalization or transfusion) outside of a surgical setting within the last year.
* Presence of coagulopathy defined as:

  * PT > 1.3 x upper limit of normal
  * PTT > 1.3 x upper limit of normal
* Uncontrolled hypothyroidism (defined as TSH below lower limit of normal). Qualifying TSH may be within 60 days prior to enrollment. If screening TSH is low, patients are eligible if free T4 is within normal limits.
* Familial bleeding diathesis
* Known diagnosis of disseminated intravascular coagulation
* Currently taking statin (i.e. rosuvastatin, atorvastatin, simvastatin) or fibrates
* Currently receiving anticoagulant therapy
* Current use of aspirin (>81 mg daily), Clopidogrel (Plavix), cilostazol (Pletal), aspirin-dipyridamole (Aggrenox).
* Known Asian descent (including Filipino, Chinese, Japanese, Korean, Vietnamese or Asian-Indian origin) due to altered metabolism of statins.
* Concomitant use of the following drugs: cyclosporine, fibrates, niacin, gemfibrozil, ketoconazole, spironolactone, cimetidine, warfarin, erythromycin, or protease inhibitors
* Known recent history of heavy alcohol use
* History of rhabdomyolysis while on statin therapy.
* Known active Hepatitis C or active Hepatitis B infection.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study due to the potential for teratogenic effects on the human fetus. Because there is an unknown but potential risk of adverse events in nursing infants secondary to the treatment of the mother with rosuvastatin, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Comparison of differences in circulating tissue factor bearing microparticles between study arms | 60 days
  Concentration of tissue factor bearing microparticles

SECONDARY OUTCOMES:
Point estimate of the rates of VTE following ovarian surgery in each study arm | 60 days
  VTE rate
Comparison of D-dimer values across study arms | 60 days
  D-dimer concentration
Compare the rates of VTE between study arms | 60 days
  VTE rate in arm A and B
Compare CRP between study arms | 60 days
  CRP concentration
Compare concentrations of TFMP, D-dimer, CRP at study timepoints. | 60 days
  Baseline vs day 60 comparison for TFMP, D-dimer, CRP on each arm
Assess incidence of major hemorrhage and clinically relevant bleeding as defined by the International Society of Thrombosis and Haemostasis | 60 days
  Major and clinically relevant non-major bleeding rates
Estimate the overall rate of any VTE | 60 days
  Overall VTE rates

CONTACTS AND LOCATIONS:
Overall Officials: Rushad Patell, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No